CLINICAL TRIAL: NCT04399564
Title: Effect of Temporary vs.Long Term Hemodialysis Catheter on Central Vein Stenosis in Long-term Hemodialysis Patients
Brief Title: Temporary vs.Long Term Hemodialysis Catheter on Central Vein Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pudong Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ShanghaiPudongH3
Record Dates: First submitted 2020-05-15; First posted 2020-05-22 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Stenosis of Arteriovenous Dialysis Fistula
Keywords: central vein stenosis; temporary hemodialysis catheters; long term hemodialysis catheter

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- temporary hemodialysis catheters (Active Comparator): one arm-temporary hemodialysis catheter
  Interventions: Device: temporary hemodialysis catheters
- long-term hemodialysis catheters (Experimental): another arm-long term hemodialysis catheter
  Interventions: Device: long-term hemodialysis catheters

INTERVENTIONS:
Device: temporary hemodialysis catheters — Vascular access using temporary vs.long-term hemodialysis catheters
  Arms: temporary hemodialysis catheters
Device: long-term hemodialysis catheters — long-term hemodialysis catheters
  Arms: long-term hemodialysis catheters

SUMMARY:
Vascular access (VA) is the most important for carrying out hemodialysis, yet it may bring in complications and leads to hemodialysis quality decline. This study aimed to explore the impact of vascular access types, including temporary vs.long term hemodialysis catheter on central vein stenosis.

DETAILED DESCRIPTION:
It is unknown whether central vein stenosis occurs after temporary or long term hemodialysis catheter in long-term hemodialysis patients. this study will aim to explore this question. Study design is randomized, controlled trial. One arm is temporary catheters in the internal jugular vein, and another arm is tunneled cuffed hemodialysis cather. 2*2 is randomly distributed.

The main outcome: central vein stenosis diagnosed by venography. The secondary outcome: the time of infection, and catheter patency. Study period: one year

ELIGIBILITY:
Inclusion Criteria:

* need to receive long-term hemodialysis no arteriovenous shunts or immature arteriovenous shunts

Exclusion Criteria:

* Uremia with heart failure or lung function failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-05-25 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
central vein stenosis | 8 weeks after temporary or long-term hemodialysis catheter
  use of venography as the primary imaging modality for vein mapping

SECONDARY OUTCOMES:
time of infection | 8 weeks
  infected in temporary or long-term hemodialysis catheters
catheter unobstructed degree | 8 weeks
  blood flow in hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Hui Min Jin, MD, Principal Investigator — Shanghai Pudong Hospital

IPD SHARING:
Plan to Share IPD: No